CLINICAL TRIAL: NCT01218750
Title: Combined Phako-Vitrectomy With ILM Peeling, Retinal Endophotocoagulation, and Intraoperative Use of Bevacizumab for Diffuse Diabetic Macular Edema
Brief Title: Triple Therapy for Diffuse Diabetic Macular Edema
Acronym: TTDDME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Department of Ophthalmology, Military Instiute of Medicine, Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46/WIM/2008
Record Dates: First submitted 2010-10-06; First posted 2010-10-11 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-09

CONDITIONS: Diffuse Diabetic Macular Edema
Keywords: DDME, ppV, ILM peeling, bevacizumab injection
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- edematous tractional epimacular membrane (Experimental): Diabatic maculopathy comes to the edematous or tractional form. It is believed that epiretinal membranes are comprised from glial components. The processes of these cells may invade through the internal limiting membrane of the retina to the vitreous causing the vitreoretinal adhesion and anomalous posterior detachment of vitreous (APVD). In the macula, APVD causes vitreo-macular traction syndrome, which results in diffuse diabetic macular edema. If vitreoschisis is present, a place of dissection is crucial. If break occurs in front of the hyalocytes remaining on the retinal surface, the vitreous layer is thick and easily shrinks concentrically, which results in the formation of epimacular membrane.
  Interventions: Procedure: Triple therapy for diffuse diabetic macular edema

INTERVENTIONS:
Procedure: Triple therapy for diffuse diabetic macular edema — Three port pars plana vitrectomy is performed by one surgeon (JR). Induction of PVD is initiated by active suction with the vitrectomy probe over the ONH and continued peripherally. Peeling of the epimacular tissue and ILM is performed by grasping the flap of the ILM with an eckhardts forceps. Trypan Blue is used to stain the ILM. Peripheral laser endophotocoagulation is performed in cases of avascular areas based on FA, active neovascularization, peripheral retinoschisis or retinal breaks. All eyes have a 1,25 mg/0,05 ml bevacizumab injection into vitreous cavity and SF6 gas tamponade at the end of the procedure. Even of absence of cataract formation, a combined procedure is performed because of exactly peripheral vitreous shaving and prevention of cataract formation.
  Other Names: Triple Therapy; Avastin (bevacizumab)

SUMMARY:
The purpose of this study is to evaluate the safety end efficacy of combined phakoemulsification and vitrectomy with retinal endophotocoagulation and intraoperative use of bevacizumab in patients with diffuse diabetic macular edema (DDME), to determine the possible preoperative and intraoperative factors that might influence surgical outcomes.

DETAILED DESCRIPTION:
The pathogenesis of the diabetic macular edema is multiple. Therefore treatment of this disease should be combined too. VEGF is involved in pathogenesis of diabetic macular edema and recently anti-VEGF agents such as bevacizumab have been shown to be beneficial in the treatment of this retinal disorder. However, endogenous VEGF is required for visual function. Growing body evidence indicates that VEGF acts also on nonvascular cells, it plays survival role on Muller cells and photoreceptors. Therefore anti-VEGF therapies should be administered with caution and not persistent. Photocoagulation in nonperfused areas eliminate increased production of VEGF, proliferation of RPE and increased production of PEDF in surrounded impact laser area. Vitrectomy with ILM peeling reliefs traction on the macula, improve oxygenation of the macula leading to decreased vascular permeability with subsequent resolution or decrease in DME. Removed ILM contains a part of the Müller cell endfeet and the horizontal gliosis. It is likely that the proliferation of GFAP-stained gliofibrils, observed in microdamaged Müller cells, preserves the blood-retinal barrier, reinforces architectural cohesion, and opposes the installation of the edema. Therefore, we made hypothesis that combined triple therapy was effective for decreasing macular thickness and improvement of vision for eyes with diffuse diabetic macular edema.

It is important for the surgeon to determine the factors that might influence surgical outcome so that patients are chosen for the procedure that they can get benefit from. Therefore, we evaluated the possible preoperative and intraoperative factors that might influence surgical outcomes

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of DDME on clinical exam, definite retinal thickening involving the center of the macula, confirmed by fluorescein angiography, with or without PVD,
2. BCVA of 0,3 or worse in log MAR units (<=70 ETDRS letter) and 1,5 or better in log MAR units (>=10 ETRDS letter),
3. mean central macular thickness greater than 250 μm on optic coherence tomography (OCT),
4. presence of vitreomacular traction or a thickened and taut posterior hyaloid or presence of an epimacular membrane.

Exclusion Criteria:

1. significant macular ischemia defined as enlarged perifoveal capillary loss (>1000 µm) by fluorescein angiography,
2. the focal macular edema due to focal leakage from microaneurysm,
3. ophthalmic disorders associated with macular edema, such as uveitis, branch or central retinal vein occlusion and pseudophakic cystoid macular edema,
4. vitreous hemorrhage or tractional retinal detachment secondary to diabetic retinopathy,
5. an ocular condition is present such that, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary abnormalities, dense subfoveal hard exudates),
6. history of retinal macular photocoagulation, intravitreal corticosteroids, or other treatment for DME within 3 months prior to enrollment,
7. history of any intraocular surgery within prior 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) and central macular thickness (CMT) | up to 1 week before surgery
  The best corrected visual acuity (BCVA) for ETDRS chart and central macular thickness (CMT) are assessed preoperatively and during the follow-up period. OCT is performed 1 mm and 6 mm diameter topography centered at the patient fixation point. We evaluate mean central retinal thickness and central retinal volume 1 mm and 6 mm in diameter.
Best-corrected visual acuity (BCVA) and central macular thickness (CMT) | 16 up to 17 weeks after surgery
  The best corrected visual acuity (BCVA) for ETDRS chart, results are converted to log MAR for statistical analysis. The central macular thickness (CMT) are assessed 1 mm diameter topography centered at the patient fixation point for OCT-SLO. We evaluate mean central retinal thickness and central retinal volume 1 mm and 6 mm in diameter.
Best-corrected visual acuity (BCVA) and central macular thickness (CMT) | 32 up to 33 weeks after surgery
  A follow-up examination include: The best corrected visual acuity (BCVA) for ETDRS chart, results are converted to log MAR for statistical analysis. The central macular thickness (CMT) are assessed 1 mm diameter topography centered at the patient fixation point for OCT-SLO. We evaluate mean central retinal thickness and central retinal volume 1 mm and 6 mm in diameter.
Best-corrected visual acuity (BCVA) and central macular thickness (CMT) | 48 up to 49 weeks after surgery
  A follow-up examination include: The best corrected visual acuity (BCVA) for ETDRS chart, results are converted to log MAR for statistical analysis. The central macular thickness (CMT) are assessed 1 mm diameter topography centered at the patient fixation point for OCT-SLO. We evaluate mean central retinal thickness and central retinal volume 1 mm and 6 mm in diameter.
Best-corrected visual acuity (BCVA) and central macular thickness (CMT) | 64 up to 65 weeks after surgery
  A follow-up examination include: The best corrected visual acuity (BCVA) for ETDRS chart, results are converted to log MAR for statistical analysis. The central macular thickness (CMT) are assessed 1 mm diameter topography centered at the patient fixation point for OCT-SLO. We evaluate mean central retinal thickness and central retinal volume 1 mm and 6 mm in diameter.

SECONDARY OUTCOMES:
Presence of vitreomacular traction or epimacular membrane, grade of DR, patients age, HbA1c level, BMI, systemic hypertension | up to 2 weeks before surgery
  The demographic characteristics of the patients including: age, grender, metabolic condition: HbA1c level, body mass index, presence of systemic hypertension, ocular condition: diabetic retinopathy stage, previous laser, presence of viteomacular traction or epiretinal membrane are recorded to eveluate the possible association with chance in postoperative BCVA.

CONTACTS AND LOCATIONS:
Overall Officials: Robaszkiewicz Jacek, dr med., Principal Investigator — Department of Ophthalmology Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Szaserów 44, Poland

REFERENCES:
- [Result] Robaszkiewicz J, Chmielewska K, Wierzbowska J, Figurska M, Frontczak-Baniewicz M, Stankiewicz A. [Combined surgical and pharmacological treatment of diabetic maculopathy]. Klin Oczna. 2010;112(1-3):19-23. Polish. PMID 20572497